CLINICAL TRIAL: NCT06710093
Title: Power of Liquid Biopsy Tracking in Immunotherapy Treated Stage IV Melanoma
Acronym: PerceIVe
Status: Not yet recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR6083
Record Dates: First submitted 2024-11-22; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Melanoma
Keywords: ctDNA testing; advanced melanoma; immune checkpoint inhibitors (ICI)
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Plasma sample, Dried Blood spot sample and Urine sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Histologically proven melanoma: Unresectable stage III or stage IV disease, with confirmed radiological disease progression within 1 month of recruitment

SUMMARY:
The advent of immune ICI has remarkably improved survival in advanced melanoma patients in the last decade. Long term responders following 2 years of treatment with immunotherapy go on to surveillance with frequent radiological imaging every 3-6 months up to 5-10 years. This not only exposes patients with a relatively low risk of recurrence to significant amounts of ionising radiation, but also increases the burden and cost on already stretched radiology departments. Therefore, this study aims to assess the feasibility and patient experience of using ctDNA with minimally invasive liquid biopsy assays as a biomarker for detecting disease relapse or progression at the point of radiological progression. Data from this pilot study will help to design a future validation study for establishing optimal liquid biopsy for surveillance in advanced melanoma patients.

DETAILED DESCRIPTION:
This prospective study will measure ctDNA in a simple plasma sample and using a dried blood spot assay, collected at the time of radiological disease progression. We will investigate the use of tumour informed and tumour naïve approaches, assessing targeted sequencing, copy number variations using whole genome low depth sequencing, fragmentomics and methylation as potential methods to improve molecular recurrence detection. We will also collect urine samples to investigate the use of cfDNA to detect relapse in the brain, which has been noted to be more challenging to detect using ctDNA in the blood than other sites of relapse.

In addition, we will investigate the use of novel immunophenotyping technology through a collaboration with MelioHealth (IMU) in the same setting. The IMU platform combines high resolution cellular analysis and machine learning to enable high-content, high-throughput and real-time cellular immunophenotyping from less than 2ml of whole blood. We hypothesize that disease relapse following immunotherapy may detectably trigger a patient's immune system memory, which may be particularly important for those patients who do not shed ctDNA.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven melanoma
* Unresectable stage III or stage IV disease, with confirmed radiological disease progression within 1 month of recruitment
* Patient has received at least 1 cycle of immunotherapy with checkpoint inhibitors for melanoma
* Undergoing standard of care active treatment with regular interval imaging or routine imaging surveillance following treatment completion/cessation
* Age over 16
* Not previously diagnosed with HIV, Hepatitis B or C (does not need testing)

Exclusion Criteria:

* Not on routine surveillance with interval imaging per standard of care
* Unable to provide informed consent due to psychological, medical or cognitive conditions.
* Unable to comply with schedule of study samples to be collected. Concurrent active malignancies needing treatment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are being enrolled from either relapsed unresectable Stage III or Stage IV melanomas
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with measurable ctDNA at the point of radiological disease progression | 1 year
  Proportion positive of ctDNA assays vs. standard imaging including CT, MRI or PET scans depending upon site of disease relapse

SECONDARY OUTCOMES:
Patient acceptance of liquid biopsy measured by proportion of enrolled patients to those invited to participate in the study | 1 year
  Patient satisfaction with using liquid biopsy for each assay measured by a question on satisfaction (Yes/No/Undecided)
Cost of standard imaging pathway and additional cost of using liquid biopsy testing | 1 year
  To assess the cost of standard imaging pathway and additional cost of using liquid biopsy testing
Proportion of patients with positive tests in the different liquid biopsy assays to detect disease relapse | 1 year
  To assess the sensitivity of different liquid biopsy assays, including plasma vs blood spot for measuring ctDNA at point of disease progression

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden, Chelsea, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Observational Pilot study, no plans to share the IPD.

REFERENCES:
- [Background] Pascual J, Attard G, Bidard FC, Curigliano G, De Mattos-Arruda L, Diehn M, Italiano A, Lindberg J, Merker JD, Montagut C, Normanno N, Pantel K, Pentheroudakis G, Popat S, Reis-Filho JS, Tie J, Seoane J, Tarazona N, Yoshino T, Turner NC. ESMO recommendations on the use of circulating tumour DNA assays for patients with cancer: a report from the ESMO Precision Medicine Working Group. Ann Oncol. 2022 Aug;33(8):750-768. doi: 10.1016/j.annonc.2022.05.520. Epub 2022 Jul 6. PMID 35809752
- [Background] Larkin J, Chiarion-Sileni V, Gonzalez R, Grob JJ, Rutkowski P, Lao CD, Cowey CL, Schadendorf D, Wagstaff J, Dummer R, Ferrucci PF, Smylie M, Hogg D, Hill A, Marquez-Rodas I, Haanen J, Guidoboni M, Maio M, Schoffski P, Carlino MS, Lebbe C, McArthur G, Ascierto PA, Daniels GA, Long GV, Bastholt L, Rizzo JI, Balogh A, Moshyk A, Hodi FS, Wolchok JD. Five-Year Survival with Combined Nivolumab and Ipilimumab in Advanced Melanoma. N Engl J Med. 2019 Oct 17;381(16):1535-1546. doi: 10.1056/NEJMoa1910836. Epub 2019 Sep 28. PMID 31562797
- [Background] Teixido C, Castillo P, Martinez-Vila C, Arance A, Alos L. Molecular Markers and Targets in Melanoma. Cells. 2021 Sep 5;10(9):2320. doi: 10.3390/cells10092320. PMID 34571969
- [Background] Lee JH, Menzies AM, Carlino MS, McEvoy AC, Sandhu S, Weppler AM, Diefenbach RJ, Dawson SJ, Kefford RF, Millward MJ, Al-Ogaili Z, Tra T, Gray ES, Wong SQ, Scolyer RA, Long GV, Rizos H. Longitudinal Monitoring of ctDNA in Patients with Melanoma and Brain Metastases Treated with Immune Checkpoint Inhibitors. Clin Cancer Res. 2020 Aug 1;26(15):4064-4071. doi: 10.1158/1078-0432.CCR-19-3926. Epub 2020 Apr 22. PMID 32321716
- [Background] Syeda MM, Wiggins JM, Corless BC, Long GV, Flaherty KT, Schadendorf D, Nathan PD, Robert C, Ribas A, Davies MA, Grob JJ, Gasal E, Squires M, Marker M, Garrett J, Brase JC, Polsky D. Circulating tumour DNA in patients with advanced melanoma treated with dabrafenib or dabrafenib plus trametinib: a clinical validation study. Lancet Oncol. 2021 Mar;22(3):370-380. doi: 10.1016/S1470-2045(20)30726-9. Epub 2021 Feb 12. PMID 33587894
- [Background] Tan L, Sandhu S, Lee RJ, Li J, Callahan J, Ftouni S, Dhomen N, Middlehurst P, Wallace A, Raleigh J, Hatzimihalis A, Henderson MA, Shackleton M, Haydon A, Mar V, Gyorki DE, Oudit D, Dawson MA, Hicks RJ, Lorigan P, McArthur GA, Marais R, Wong SQ, Dawson SJ. Prediction and monitoring of relapse in stage III melanoma using circulating tumor DNA. Ann Oncol. 2019 May 1;30(5):804-814. doi: 10.1093/annonc/mdz048. PMID 30838379
- [Background] Lee RJ, Gremel G, Marshall A, Myers KA, Fisher N, Dunn JA, Dhomen N, Corrie PG, Middleton MR, Lorigan P, Marais R. Circulating tumor DNA predicts survival in patients with resected high-risk stage II/III melanoma. Ann Oncol. 2018 Feb 1;29(2):490-496. doi: 10.1093/annonc/mdx717. PMID 29112704
- [Background] MANDEL P, METAIS P. [Nuclear Acids In Human Blood Plasma]. C R Seances Soc Biol Fil. 1948 Feb;142(3-4):241-3. No abstract available. French. PMID 18875018
- [Background] Tan AC, Emmett L, Lo S, Liu V, Kapoor R, Carlino MS, Guminski AD, Long GV, Menzies AM. FDG-PET response and outcome from anti-PD-1 therapy in metastatic melanoma. Ann Oncol. 2018 Oct 1;29(10):2115-2120. doi: 10.1093/annonc/mdy330. PMID 30137228
- [Background] Eroglu Z, Krinshpun S, Kalashnikova E, Sudhaman S, Ozturk Topcu T, Nichols M, Martin J, Bui KM, Palsuledesai CC, Malhotra M, Olshan P, Markowitz J, Khushalani NI, Tarhini AA, Messina JL, Aleshin A. Circulating tumor DNA-based molecular residual disease detection for treatment monitoring in advanced melanoma patients. Cancer. 2023 Jun 1;129(11):1723-1734. doi: 10.1002/cncr.34716. Epub 2023 Mar 4. PMID 36869646
- See also: Recommendations | Melanoma: assessment and management | Guidance | NICE — https://www.nice.org.uk/guidance/ng14/chapter/Recommendations#follow-up-after-treatment-for-melanoma